CLINICAL TRIAL: NCT00779038
Title: Clinical Outcome Study in Postoperative Pain Management to Demonstrate the Efficacy and Safety of IONSYS (Fentanyl ITS Iontophoretic Transdermal System) in Daily Clinical Practice and to Assess Its Convenience (IPAC)
Brief Title: Safety and Efficacy Study of Fentanyl Iontophoretic Transdermal System (ITS) for Management of Moderate to Severe Acute Pain in Participants Who Have Undergone Elective Spine or Orthopedic Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped prematurely in 2008 due to IONSYS withdrawal off the market globally
Sponsor: Janssen Cilag N.V./S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015121; FENHYDPAI4014; 2008-002074-35
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2013-02-13 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Pain, Postoperative
Keywords: IONSYS; Fentanyl Iontophoretic Transdermal System; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fentanyl ITS (Experimental): 40 microgram (mcg) per 10 minutes of fentanyl dose up to a maximum of 240 mcg (6 doses each of 10 minutes duration) per hour but not more than a maximum of 3.2 milligram (80 doses) within a 24 hour period from an Iontophoretic Transdermal System (ITS). Total duration of treatment will be 72 hours.
  Interventions: Drug: Fentanyl ITS

INTERVENTIONS:
Drug: Fentanyl ITS — 40 mcg per 10 minutes of fentanyl dose up to a maximum of 240 mcg (6 doses each of 10 minutes duration) per hour but not more than a maximum of 3.2 milligram (80 doses) within a 24 hour period from an ITS. Total duration of treatment will be 72 hours.
  Other Names: IONSYS

SUMMARY:
The purpose of this study is to evaluate in daily clinical practice the safety and efficacy of fentanyl Iontophoretic Transdermal (through the skin) System (ITS) for management of moderate (medium level of seriousness) to severe (very serious) acute (a quick and severe) pain in participants who have undergone elective spine or orthopedic (related to bones) surgery.

DETAILED DESCRIPTION:
This is an open-label (participants and physicians are told which treatment the participants are receiving), multi-center (when more than one hospital or medical school team work on a medical research study), single-arm study of fentanyl ITS. The study will consist of 2 phases: screening phase and an open-label treatment phase. The duration of participation in the study for an individual participant will be 72 hours. All eligible participants (who require pain treatment with strong opioids [morphine like medications] for at least 48 hours after an elective spine or elective orthopedic surgery) will be treated with fentanyl ITS, delivering 40 microgram (mcg) fentanyl per on-demand dose, each deliver over 10 minutes for a maximum of 6 doses per hour (240 mcg per hour) for 24 hours or a maximum of 80 doses (3.2 milligram). Participants will be analyzed for the use of intravenous (giving a medicine directly into a vein) access during postoperative pain treatment with fentanyl ITS. Participant's safety will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Participants who will undergo elective spine or orthopedic (related to bones) surgery
* Participants who are expected to have moderate (medium level of seriousness) or severe (very serious) pain requiring parenteral (given by injection) opioids (morphine like medications) for at least 48 hours after surgery
* Participants who have been admitted to the Post Anesthesia Care Unit (PACU) after general anesthesia, spinal anesthetic of less than 4 hours duration of action or epidural (outside the spinal cord) anesthesia
* Participants who are alert and breathing spontaneously for at least 30 minutes in the PACU
* Participants with a pain score less than or equal to 4 out of 10 on a Numerical Rating Scale (NRS) at movement of the operated limb or body region, after titration to comfort according to current postoperative procedures

Exclusion Criteria:

* Participants with active systemic skin disease or active local skin disease that prohibit fentanyl Iontophoretic Transdermal (through the skin) System (ITS) application
* Participants with a history of allergy or hypersensitivity to fentanyl and/or an allergy/hypersensitivity to skin adhesives and/or cetylpyridinium chloride
* Participants who received regular treatment with transdermal strong opioids within 14 days prior to surgery
* Participants who are known or suspected to have abused any drug substance or alcohol
* Participants who will probably require additional surgical procedures within 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag N.V./S.A., Belgium Clinical Trial, Study Director — Janssen Cilag N.V./S.A.
Locations (3):
- Belgium (3):
  - Aalst
  - Brussels
  - Edegem

RESULTS

PARTICIPANT FLOW:
Groups:
- Fentanyl ITS: Participants received 40 microgram (mcg) per 10 minutes of fentanyl dose up to a maximum of 240 mcg (6 doses each of 10 minutes duration) per hour but not more than a maximum of 3.2 milligram (80 doses) within a 24 hour period from an Iontophoretic Transdermal System (ITS [a device which uses an electric current to move drug through the skin into the blood]), applied on the intact, non-irritated skin on the chest or upper arm. Duration of study treatment was 72 hours.
Period: Overall Study
Arm/Group | Fentanyl ITS
Started | 13
Completed | 0
Not Completed | 13
Not completed — Study Prematurely Terminated | 13

BASELINE CHARACTERISTICS:
Groups:
- Fentanyl ITS: Participants received 40 microgram (mcg) per 10 minutes of fentanyl dose up to a maximum of 240 mcg (6 doses each of 10 minutes duration) per hour but not more than a maximum of 3.2 milligram (80 doses) within a 24 hour period from an Iontophoretic Transdermal System (ITS), applied on the intact, non-irritated skin on the chest or upper arm. Duration of study treatment was 72 hours.
Arm/Group | Fentanyl ITS
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Intravenous Administration During Treatment With Fentanyl Iontophoretic Transdermal System (ITS) at Hour 24
Description: Total number of participants who required intravenous administration (when medicine is given directly into a vein) postoperatively, for treating study treatment related side effect or for additional pain control, during treatment with fentanyl ITS was assessed.
Time Frame: Hour 24
Population: Data was not analyzed because there were insufficient participants to perform a meaningful efficacy analysis due to premature study termination.
Arm/Group | Fentanyl ITS
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Patient Global Assessment (PGA) of Method of Pain Control
Description: The PGA was based on categorical evaluation (poor, fair, good or excellent) for the method of pain control by asking following question from the participants: "Overall, would you rate this method of pain control as being poor, fair, good, or excellent?"
Time Frame: Hour 72 or early withdrawal
Population: as for outcome 1
Arm/Group | Fentanyl ITS
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Nurse Global Assessment of Method of Pain Control
Description: The nurse global assessment was based on categorical evaluation (poor, fair, good or excellent) for the method of pain control by asking following question from the nurses: "Overall, would you rate this method of pain control as being poor, fair, good, or excellent?"
Time Frame: Hour 72 or early withdrawal
Population: as for outcome 1
Arm/Group | Fentanyl ITS
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Physician Global Assessment of Method of Pain Control
Description: The physician global assessment was based on categorical evaluation (poor, fair, good or excellent) for the method of pain control by asking following question from the Physicians: "Overall, would you rate this method of pain control as being poor, fair, good, or excellent?"
Time Frame: Hour 72 or early withdrawal
Population: as for outcome 1
Arm/Group | Fentanyl ITS
Number analyzed (Participants) | 0

5. Primary Outcome: Number of Participants With Intravenous Administration During Treatment With Fentanyl ITS at Hour 48
Description: Total number of participants who required intravenous administration postoperatively, for treating study treatment related side effect or for additional pain control, during treatment with fentanyl ITS was assessed.
Time Frame: Hour 48
Population: as for outcome 1
Arm/Group | Fentanyl ITS
Number analyzed (Participants) | 0

6. Primary Outcome: Number of Participants With Intravenous Administration During Treatment With Fentanyl ITS at End of Study Treatment
Description: as for outcome 5
Time Frame: End of Study treatment (Hour 72)
Population: as for outcome 1
Arm/Group | Fentanyl ITS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment upto Day 14
Arm/Group | Fentanyl ITS
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl ITS (N=13)
Peroneal nerve palsy (severe) (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fentanyl ITS (N=13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Application site reaction (General disorders) | 2
Application site discolouration (General disorders) | 1 (2)
Application site swelling (General disorders) | 1
Application site pruritus (left side) (General disorders) | 1
Application site pruritus (right side) (General disorders) | 1
Euphoric mood (Psychiatric disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 1
Inadequate analgesia (Injury, poisoning and procedural complications) | 2
Peroneal nerve palsy (moderate) (Nervous system disorders) | 1
Pyrexia (General disorders) | 1
Urinary retension (Renal and urinary disorders) | 3
Application site reaction (left side) (General disorders) | 1
Application site reaction (right side) (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
No efficacy results were reported because the study was prematurely terminated, following the worldwide voluntary withdrawal of Fentanyl Iontophoretic Transdermal System (IONSYS) by Janssen-Cilag.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No